CLINICAL TRIAL: NCT00691548
Title: Non Invasive Imaging of Cetuximab-Zirconium-89 Uptake With PET: a Phase I Trial in Stage IV Cancer
Brief Title: Non-invasive Imaging of Cetuximab-Zr. 89 Uptake Wit PET: a Phase I Trial in Stage IV Cancer Patients
Acronym: Cetuximab Zr89
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cetuximab-Zr.89 fase I; 08-3-039 (MEC)
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Stage IV Cancer
Keywords: Stage IV cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Cetuximab-Zr. 89

INTERVENTIONS:
Drug: Cetuximab-Zr. 89 — Step 1: Determination of the toxicity of two low doses of 89Zr-cetuximab In three patients a standard loading dose of 400 mg/m2 of cetuximab will be administered, partly labelled with 89Zr (60 MBq, 2.5mg) on day 0.
  On day 14, a second injection with dose of 250 mg/m2 of cetuximab, partly labelled with 89Zr (60 MBq, 2.5mg), will be given.
  Step 2: Determination of the toxicity of one larger dose of 89Zr-cetuximab A standard loading dose of 400 mg/m2 of cetuximab will be administered in 3 patients, a part labelled with 89Zr (120MBq, 5mg).

SUMMARY:
Non invasive imaging of cetuximab uptake with PET could help to select the patients who could be treated by cetuximab, a registered but expensive monoclonal antibody against EGFR. Other monoclonal antibodies labelled with Zirconium-89 have already been used with success in patients. The combination of cetuximab labelled with Zirconium-89 is a promising new probe to determine cetuximab uptake, which has been tested in various pre-clinical animal models in Maastricht with excellent results.

We propose a two step study design (see figure 1). As our ultimate goal for the future is to determine the uptake of 89Zr-cetuximab in the tumour before and during therapy, we need to investigate the toxicity of two consecutive low doses of 89Zr-cetuximab in the first place. However, as in future studies and in some patients, it is also possible that a single, larger dose of 89Zr-cetuximab is needed to obtain the best image quality, we will also investigate the toxicity of a single larger dose.

Step 1: Determination of the toxicity of two low doses of 89Zr-cetuximab In three patients a standard loading dose of 400 mg/m2 of cetuximab will be administered, partly labelled with 89Zr (60 MBq, 2.5mg) on day 0.

On day 14, a second injection with dose of 250 mg/m2 of cetuximab, partly labelled with 89Zr (60 MBq, 2.5mg), will be given.

Step 2: Determination of the toxicity of one larger dose of 89Zr-cetuximab A standard loading dose of 400 mg/m2 of cetuximab will be administered in 3 patients, a part labelled with 89Zr (120MBq, 5mg).

DETAILED DESCRIPTION:
Toxicity will be scored twice a week from the day of first injection (day 0) up to day 14, according to the CTCAE3.0 scoring system. As after 14 days, the activity of Zr89 is low (four half-lives of Zr89 is 4 x 3.2 days = 12.8 days), no additional toxic effect is expected. Blood sampling will be done weekly (haematology, liver and kidney function).

When in 0/3 patients a toxicity of grade 3 or more has occurred step 2 is considered safe. If in 1/3 patients a grade 3 has occurred, 3 more patients will be included in this step. If another grade 3 toxicity occurs in 1/3 patients, the study will be stopped. When at maximum 1/6 patients experience a grade 3 toxicity, this step will be considered safe. When step 2 is considered safe, the study is ended.

After the injection, visualization of all tumour sites will be analyzed by performing a PET-CT scan on day 4, 5 and 6 post injection. An additional scan on day 3 or 7 is optional.* At day 5 post injection a perfusion PET-CT will be performed.

ELIGIBILITY:
Inclusion criteria:

* Stage IV cancer (primary or recurrent)
* Normal white blood cell count and formula
* Normal platelet count
* No anemia requiring blood transfusion or erythropoietin
* Adequate hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution).
* Calculated Creatinin clearance at least 60 ml/min
* No previous administration of cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Toxicity (CTCAE 3.0) | 2 weeks

SECONDARY OUTCOMES:
Image Quality (Tumour-to-Background Ratio) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, Dr., Principal Investigator — Maastro Radiation Oncology
Locations (1):
- Maastro Clinic, Maastricht, Netherlands